CLINICAL TRIAL: NCT03710291
Title: A Phase 3b, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of TRC101 in Delaying Chronic Kidney Disease Progression in Subjects With Metabolic Acidosis
Brief Title: Evaluation of Effect of TRC101 on Progression of Chronic Kidney Disease in Subjects With Metabolic Acidosis
Acronym: VALOR-CKD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: Tricida, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRCA-303; 2018-001303-36 (EudraCT Number)
Record Dates: First submitted 2018-10-11; First posted 2018-10-18 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Metabolic Acidosis; Chronic Kidney Disease
Keywords: serum bicarbonate; renal outcomes; TRC101; eGFR; veverimer
MeSH Terms: conditions — Acidosis; Renal Insufficiency, Chronic | interventions — veverimer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TRC101 (Experimental)
  Interventions: Drug: TRC101
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRC101 — Oral, non-absorbed, polymeric hydrochloric acid binder
  Other Names: Veverimer
  Arms: TRC101
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of TRC101 on the progression of chronic kidney disease (CKD) and to evaluate the safety profile of TRC101 in CKD patients with metabolic acidosis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial. Eligible subjects will be randomized in a 1:1 ratio to TRC101 or placebo. The primary endpoint of the study will be progression of renal disease, defined by time to first occurrence of any event in the composite endpoint consisting of a confirmed ≥ 40% reduction in eGFR, end-stage renal disease (ESRD), and renal death. The study will terminate when the independent blinded Clinical Endpoint Adjudication Committee has positively adjudicated the targeted number of primary efficacy endpoint events. The maximum duration of follow-up for a randomized subject is anticipated to be approximately 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Estimated glomerular filtration rate (eGFR) 20 - 40 mL/min/1.73m^2.
* Serum bicarbonate 12 - 20 mEq/L.
* On maximum tolerated dose of ACE inhibitor and/or ARB.

Exclusion Criteria:

* Acute metabolic acidosis.
* Anticipated dialysis or kidney transplant within 6 months.
* Recent acute kidney injury.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1480 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Progression of chronic kidney disease | Through study completion, up to approximately 6 years.
  Time to first occurrence of: a confirmed ≥40% reduction in eGFR; ESRD; renal death.

SECONDARY OUTCOMES:
Death (all-cause), ESRD or a confirmed ≥50% reduction in eGFR | Through study completion, up to approximately 6 years.
  Time to first occurrence of: death (all-cause); ESRD; a confirmed ≥50% reduction in eGFR.
Physical functioning (subjective) | 18 months after randomization.
  Kidney Disease Quality of Life Physical Functioning Survey.
Physical functioning (objective) | 18 months after randomization.
  Repeated chair stand test.
ESRD or renal death | Through study completion, up to approximately 6 years.
  Time to ESRD or renal death.
Primary outcome measure OR cardiovascular death | Through study completion, up to approximately 6 years.
  Time to first occurrence of: a confirmed ≥40% reduction in eGFR; ESRD; renal death; cardiovascular death.
Serum creatinine | Through study completion, up to approximately 6 years.
  Time to first occurrence of a confirmed doubling of serum creatinine.
≥50% reduction in eGFR | Through study completion, up to approximately 6 years.
  Time to first occurrence of a confirmed ≥50% reduction in eGFR.
≥40% reduction in eGFR | Through study completion, up to approximately 6 years.
  Time to first occurrence of a confirmed ≥40% reduction in eGFR.
All-cause hospitalization | Through study completion, up to approximately 6 years.
  Frequency of all-cause hospitalization.
Cardiovascular death | Through study completion, up to approximately 6 years.
  Time to cardiovascular death.
All-cause mortality | Through study completion, up to approximately 6 years.
  Time to all-cause mortality.

OTHER OUTCOMES:
Safety of TRC101 | Through study completion, up to approximately 6 years.
  Frequency, intensity, and relationship to study drug of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Locations (203):
- United States (20):
  - Investigative Site 4136, Azusa, California
  - Investigative Site 4148, Denver, Colorado
  - Investigative Site 4157, Boca Raton, Florida
  - Investigative Site 4146, Bradenton, Florida
  - Investigative Site 4102, Coral Springs, Florida
  - Investigative Site 4153, Fort Lauderdale, Florida
  - Investigative Site 4122, Hollywood, Florida
  - Investigative Site 4123, Hollywood, Florida
  - Investigative Site 4104, Miami, Florida
  - Investigative Site 4130, Miami Lakes, Florida
  - Investigative Site 4116, Port Charlotte, Florida
  - Investigative Site 4152, Tampa, Florida
  - Investigative Site 4127, Augusta, Georgia
  - Investigative Site 4141, Greenbelt, Maryland
  - Investigative Site 4155, Kansas City, Missouri
  - Investigative Site 4108, Greenville, North Carolina
  - Investigative Site 4106, Kinston, North Carolina
  - Investigative Site 4107, New Bern, North Carolina
  - Investigative Site 4124, Bethlehem, Pennsylvania
  - Investigative Site 4132, Nashville, Tennessee
- Albania (2):
  - Investigative Site 1103, Shkodër
  - Investigative Site 1101, Tirana
- Argentina (6):
  - Investigative Site 4402, Buenos Aires
  - Investigative Site 4410, Corrientes
  - Investigative Site 4414, Córdoba
  - Investigative Site 4408, Córdoba
  - Investigative Site 4405, Mar del Plata
  - Investigative Site 4409, San Luis
- Armenia (6):
  - Investigative Site 2803, Yerevan
  - Investigative Site 2809, Yerevan
  - Investigative Site 2802, Yerevan
  - Investigative site 2801, Yerevan
  - Investigative Site 2805, Yerevan
  - Investigative Site 2807, Yerevan
- Investigative Site 5101, Gosford, Australia
- Investigative Site 1502, Grodno, Belarus
- Belgium (2):
  - Investigative Site 3108, Liège
  - Investigative Site 3103, Liège
- Brazil (9):
  - Investigative Site 4518, Caxias do Sul
  - Investigative Site 4516, Curitiba
  - Investigative Site 4504, Curitiba
  - Investigative Site 4507, Juiz de Fora
  - Investigative Site 4517, São Paulo
  - Investigative Site 4508, São Paulo
  - Investigative Site 4509, São Paulo
  - Investigative Site 4506, São Paulo
  - Investigative Site 4519, São Paulo
- Bulgaria (10):
  - Investigative Site 1211, Kozloduy
  - Investigative Site 1213, Montana
  - Investigative Site 1210, Pleven
  - Investigative Site 1205, Rousse
  - Investigative Site 1212, Rousse
  - Investigative Site 1206, Sevlievo
  - Investigative Site 1204, Sliven
  - Investigative Site 1201, Sofia
  - Investigative Site 1208, Veliko Tarnovo
  - Investigative Site 1203, Yambol
- Canada (5):
  - Investigative Site 4203, Brampton
  - Investigative Site 4202, Kitchener
  - Investigative Site 4201, London
  - Investigative Site 4204, Québec
  - Investigative Site 4208, Winnipeg
- Chile (3):
  - Investigative Site 4604, Concepción
  - Investigative Site 4601, Providencia
  - Investigative Site 4602, Temuco
- Colombia (5):
  - Investigative Site 4703, Barranquilla
  - Investigative Site 4708, Barranquilla
  - Investigative Site 4712, Barranquilla
  - Investigative Site 4705, Cali
  - Investigative Site 4709, Zipaquirá
- Czechia (2):
  - Investigative Site 2106, Sokolov
  - Investigative Site 2107, Znojmo
- France (2):
  - Investigative Site 3209, Boulogne-Billancourt
  - Investigative Site 3205, Lille
- Georgia (13):
  - Investigative Site 2201, Batumi
  - Investigative Site 2202, Kutaisi
  - Investigative Site 2208, Tbilisi
  - Investigative Site 2205, Tbilisi
  - Investigative Site 2211, Tbilisi
  - Investigative Site 2204, Tbilisi
  - Investigative Site 2206, Tbilisi
  - Investigative Site 2207, Tbilisi
  - Investigative Site 2209, Tbilisi
  - Investigative Site 2212, Tbilisi
  - Investigative Site 2213, Tbilisi
  - Investigative Site 2214, Tbilisi
  - Investigative Site 2210, Tbilisi
- Hong Kong (4):
  - Investigative Site 6101, Hong Kong
  - Investigative Site 6103, Hong Kong
  - Investigative Site 6105, Hong Kong
  - Investigative Site 6104, Shatin
- Hungary (7):
  - Investigative Site 2311, Baja
  - Investigative Site 2312, Budapest
  - Investigative Site 2304, Budapest
  - Investigative Site 2306, Győr
  - Investigative Site 2309, Kaposvár
  - Investigative Site 2310, Kistarcsa
  - Investigative Site 2316, Nagykanizsa
- Israel (5):
  - Investigative Site 3913, Afula
  - Investigative Site 3902, Ashkelon
  - Investigative Site 3905, Jerusalem
  - Investigative Site 3911, Tel Aviv
  - Investigative Site 3903, Tiberias
- Italy (6):
  - Investigative Site 3408, Genova
  - Investigative Site 3407, Messina
  - Investigative Site 3405, Milan
  - Investigative Site 3406, Napoli
  - Investigative Site 3402, Pavia
  - Investigative Site 3409, Reggio Calabria
- Malaysia (9):
  - Investigative Site 6208, Klang
  - Investigative Site 6203, Kota Bharu
  - Investigative Site 6207, Kota Bharu
  - Investigative Site 6202, Kuala Lumpur
  - Investigative Site 6204, Kuantan
  - Investigative Site 6205, Kulim
  - Investigative Site 6210, Pulau Pinang
  - Investigative Site 6206, Seri Manjung
  - Investigative Site 6201, Sungai Petani
- Mexico (15):
  - Investigative Site 4307, Cuernavaca
  - Investigative Site 4313, Guadalajara
  - Investigative Site 4304, Guadalajara
  - Investigative Site 4319, Guadalajara
  - Investigative Site 4325, Mexico City
  - Investigative Site 4311, Mexico City
  - Investigative Site 4302, Mexico City
  - Investigative Site 4316, Mérida
  - Investigative Site 4301, Mérida
  - Investigative Site 4320, Monterrey
  - Investigative Site 4315, Morelia
  - Investigative Site 4324, Morelia
  - Investigative Site 4310, Veracruz
  - Investigative Site 4305, Xalapa
  - Investigative Site 4312, Zapopan
- Netherlands (3):
  - Investigative Site 3507, Alkmaar
  - Investigative Site 3505, Amersfoort
  - Investigative Site 3503, Groningen
- North Macedonia (5):
  - Investigative Site 1304, Bitola
  - Investigative Site 1305, Shtip
  - Investigative Site 1301, Skopje
  - Investigative Site 1303, Skopje
  - Investigative Site 1302, Struga
- Poland (3):
  - Investigative Site 2421, Krakow
  - Investigative Site 2414, Warsaw
  - Investigative Site 2412, Zabrze
- Portugal (4):
  - Investigative Site 3604, Aveiro
  - Investigative Site 3603, Lisbon
  - Investigative Site 3607, Lisbon
  - Investigative Site 3605, Vila Nova de Gaia
- Investigative Site 1412, Oradea, Romania
- Serbia (7):
  - Investigative Site 2501, Belgrade
  - Investigative Site 2508, Kragujevac
  - Investigative Site 2510, Kruševac
  - Investigative Site 2505, Niš
  - Investigative Site 2514, Užice
  - Investigative Site 2503, Vršac
  - Investigative Site 2511, Zaječar
- Singapore (3):
  - Investigative Site 6401, Singapore
  - Investigative Site 6403, Singapore
  - Investigative Site 6404, Singapore
- Slovakia (3):
  - Investigative Site 2604, Košice
  - Investigative Site 2606, Košice
  - Investigative Site 2603, Svidník
- South Korea (9):
  - Investigative Site 5207, Ansan
  - Investigative Site 5203, Anyang
  - Investigative Site 5218, Cheonan
  - Investigative Site 5204, Daejeon
  - Investigative Site 5205, Goyang
  - Investigative Site 5215, Guri-si
  - Investigative Site 5213, Seoul
  - Investigative Site 5208, Seoul
  - Investigative Site 5212, Wŏnju
- Spain (3):
  - Investigative Site 3716, Barcelona
  - Investigative Site 3707, Barcelona
  - Investigative Site 3706, Barcelona
- Taiwan (10):
  - Investigative Site 6512, Changhua
  - Investigative Site 6502, Hualien City
  - Investigative Site 6501, Kaohsiung City
  - Investigative Site 6504, New Taipei City
  - Investigative Site 6506, Taichung
  - Investigative Site 6510, Taichung
  - Investigative Site 6507, Taichung
  - Investigative Site 6503, Tainan
  - Investigative Site 6509, Taipei
  - Investigative Site 6511, Taipei
- Ukraine (16):
  - Investigative Site 2712, Dnipro
  - Investigative Site 2714, Ivano-Frankivsk
  - Investigative Site 2717, Kharkiv
  - Investigative Site 2713, Kharkiv
  - Investigative Site 2721, Kharkiv
  - Investigative Site 2704, Kharkiv
  - Investigative Site 2707, Kharkiv
  - Investigative Site 2706, Kyiv
  - Investigative Site 2703, Kyiv
  - Investigative Site 2709, Kyiv
  - Investigative Site 2705, Kyiv
  - Investigative Site 2710, Kyiv
  - Investigative Site 2716, Kyiv
  - Investigative Site 2718, Ternopil
  - Investigative Site 2719, Zaporizhzhya
  - Investigative Site 2715, Zhytomyr
- United Kingdom (3):
  - Investigative Site 3815, Coventry
  - Investigative Site 3804, Nottingham
  - Investigative Site 3801, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tangri N, Mathur VS, Bushinsky DA, Klaerner G, Li E, Parsell D, Stasiv Y, Walker M, Wesson DE, Wheeler DC, Perkovic V, Inker LA. VALOR-CKD: A Multicenter, Randomized, Double-Blind Placebo-Controlled Trial Evaluating Veverimer in Slowing Progression of CKD in Patients with Metabolic Acidosis. J Am Soc Nephrol. 2024 Mar 1;35(3):311-320. doi: 10.1681/ASN.0000000000000292. Epub 2024 Jan 23. PMID 38261535
- [Derived] Hultin S, Johnson DW, Badve SV. Recent evidence on the effect of treatment of metabolic acid on the progression of kidney disease. Curr Opin Nephrol Hypertens. 2021 Sep 1;30(5):467-473. doi: 10.1097/MNH.0000000000000728. PMID 34009141